CLINICAL TRIAL: NCT03365544
Title: The Effect of Different Time-restricted Eating Windows on Body Composition
Brief Title: Effect of Eating Timing on Body Composition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, Professor of School of Kinesiology, Western University, Canada
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110492
Record Dates: First submitted 2017-11-27; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Time-Restricted Eating (16:8); Fasting
MeSH Terms: conditions — Intermittent Fasting; Fasting

STUDY DESIGN:
Intervention Model Description: One group has their eating window between 6am-2pm and the other has their eating window between 2pm-10pm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6am-2pm eating window (Experimental): 4 weeks of time restricted eating between 6am-2pm.
  Interventions: Other: Time-restricted eating
- 2pm-10pm eating window (Experimental): 4 weeks of time restricted eating between 2pm-10pm.
  Interventions: Other: Time-restricted eating

INTERVENTIONS:
Other: Time-restricted eating — Groups will be required to only ingest calories in their designated 8 hour eating window.
  Other Names: Intermittent Fasting

SUMMARY:
This study will examine the effect of eating timing on body composition. Previous studies have shown that restricting food intake to 8 hours a day can result in losses in body fat and an up-regulation of fat use. The purpose of this study is to assess changes in body composition when the eating window time is from 6am-2pm vs 2pm-10pm.

Hypothesis: The 2-10pm eating window will result in significantly greater changes in body composition (i.e. decreased fat mass) and the 2pm-10pm window will result in better adherence.

Methods: Body composition (fat and lean mass) will be assessed by air displacement densitometry (Bod Pod). Measures will be made over 4 weeks (pre-) and (post) dietary treatment. Adherence will also be assessed by a questionnaire to determine the ease/difficulty of the treatment.

DETAILED DESCRIPTION:
Purpose The purpose of the study is to determine whether the eating window of a time-restricted eating protocol affects changes in body composition. It is hypothesized that the afternoon group will have better adherence to their experimental protocol and have greater changes in body composition.

Sample The sample will include 20 healthy adult participants ranging in age from 18-25 that volunteer to participate in the study. Participants will be required to have a body mass index above 26 (BMI=weight(kg)/height(m)2). All individuals must give written informed consent in order to participate in the study. Exclusion criteria include a history of intermittent fasting in the past 6 months, diabetes, or pregnancy and BMI less than 25.9.

Procedure Inclusion/exclusion criteria will be explicitly stated throughout the recruitment process. Potential participants will be recruited through advertising using posters placed through the University of Westerns campus as well as via presentations in classrooms (using the information from the advertising flyers). Individuals who email Bryce Knapp will be invited to a meeting to discuss the study. After the evaluation and information meeting, the individual will be given up to 3 days to determine if they want to participate and give their informed consent. See attached form in the consent section of the ethics application.

Measurement: All individuals will have their body composition measured. Body composition will be measured using air displacement densitometry "Bod Pod". Measurements will be taken twice prior to the intervention and twice on successive days post-intervention. Individuals will also be asked to fill out a biweekly modified dialysis diet and fluid non-adherence questionnaires (DDFQ) with added checkboxes to record which days they complied with the required protocol and 2 questions regarding any struggles the participants experienced. This will be used to assess the adherence to the protocols.

Protocol: 20 participants matched for BMI will be assigned to one of two groups. The two groups will be assigned an eating period of 6am-2pm or 2pm-10pm and instructed not to ingest calories outside of their respective eating window. The interventions will last 4 weeks with individuals being asked to comply to their eating window a minimum of 5 days per week. This will be measured using the modified DDFQ. All testing will be completed by Bryce Knapp under the supervision of Dr. Lemon. The changes in fat mass will be analyzed using a 2-way ANOVA and the adherence will be measured using an independent t-test.

ELIGIBILITY:
Inclusion Criteria:

* 18-25 years of age
* men and women

Exclusion Criteria:

* Body mass index less than 26
* No history of intermittent fasting in the past 6 months
* No participants with diabetes
* Are pregnant or become pregnant (self-reported)
* Have symptoms or take medication for a respiratory, cardiovascular, neuromuscular, or metabolic disease

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change in Fat mass using "Bod Pod" | 4 weeks
  Measuring the change in fat mass between the two groups using air displacement densitometry "Bod Pod"

SECONDARY OUTCOMES:
Adherence using the dialysis diet and fluid non-adherence questionnaire. | 4 weeks
  Measuring adherence of the two groups using the DDFQ non adherence questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lemon, PhD, Principal Investigator — Western University, Canada
Locations (1):
- Exercise Nutrition Laboratory (Western University), London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moro T, Tinsley G, Bianco A, Marcolin G, Pacelli QF, Battaglia G, Palma A, Gentil P, Neri M, Paoli A. Effects of eight weeks of time-restricted feeding (16/8) on basal metabolism, maximal strength, body composition, inflammation, and cardiovascular risk factors in resistance-trained males. J Transl Med. 2016 Oct 13;14(1):290. doi: 10.1186/s12967-016-1044-0. PMID 27737674
- [Background] Rothschild J, Hoddy KK, Jambazian P, Varady KA. Time-restricted feeding and risk of metabolic disease: a review of human and animal studies. Nutr Rev. 2014 May;72(5):308-18. doi: 10.1111/nure.12104. Epub 2014 Apr 16. PMID 24739093
- [Background] Tinsley GM, La Bounty PM. Effects of intermittent fasting on body composition and clinical health markers in humans. Nutr Rev. 2015 Oct;73(10):661-74. doi: 10.1093/nutrit/nuv041. Epub 2015 Sep 15. PMID 26374764

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT03365544/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT03365544/ICF_001.pdf